CLINICAL TRIAL: NCT01082354
Title: Non Interventional Study on the Follow-up, by Specialists, of Short Children Born Small for Gestational Age and Treated With SAIZEN®- SEPAGE Study
Brief Title: A Pharmaco-epidemiological Study of Short Patients Born Small for Gestational Age (SGA), Treated With Saizen® (Recombinant Somatropin)
Acronym: SEPAGE
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A.S, France (Industry)
Responsible Party: Sponsor
Other Study IDs: IMP28018
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Infant, Small for Gestational Age
Keywords: Infant, Low birth weight; Infant, Low birth height; Infant, Small for Gestational Age
MeSH Terms: interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: recombinant somatropin — as per standard practice
  Other Names: Saizen

SUMMARY:
This one-arm, multi-centric, non-randomized, observational, open label, prospective study was designed to study short subjects born SGA, by pediatricians, endocrinologists or physicians in private, mixed private and hospital practice treated with Saizen.

DETAILED DESCRIPTION:
The term "small for gestational age" (SGA) is a pathological medical condition known since about two decades supported by two consensus conferences of 2001. It inhibits the height and/or weight of the child at birth without prejudging the mechanisms that alter these. This study will be carried out by hospital pediatricians, endocrinologists or physicians in private, mixed private and hospital practice in metropolitan France. Subjects will be monitored by doctors in accordance with the normal scope of follow-up of pathology until their final growth and until they reach adult height and/or until the treatment is discontinued. The participating doctors will include all the short SGA subjects coming for consultation or the follow-up (for less than 12 months) of their treatment by Saizen in this study. The inclusions will take place over a period of 21 months.

OBJECTIVES

Primary objective:

* To describe the characteristics of short children born SGA (SGA subjects) treated with Saizen

Secondary objectives:

* To describe the terms and conditions for the prescription of Saizen in terms of dosage, duration of treatment, reason for discontinuation and compliance
* To describe the effects of Saizen on growth and final height
* To describe the tolerance of Saizen. For each subject and during each visit, the participating doctor will complete an electronic data collection form.

ELIGIBILITY:
Inclusion Criteria:

* Short children born SGA requiring treatment with Saizen, new to growth hormone treatment or being treated with growth hormones for less than 12 months of inclusion
* Subjects whose parents have given their written consent for participation in this study

Exclusion Criteria:

* Contra-indication in the treatment with Saizen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 48 hospital pediatric and endocrinology centers or in mixed private and hospital practice will enroll 150 children
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Auxological characteristics (height and weight, head circumference, growth curve used, bone age) and Clinical examination (cardiac frequency, systolic blood pressure, diastolic blood pressure, Tanner pubertal stage) | Inclusion visit to follow-up visits at 3, 6 and 12 month and annual until the adult height is reached and or the final discontinuation of the treatment
Saizen prescription and compliance to treatment | Inclusion visit to follow-up visits at 3, 6 and 12 month and annual until the adult height is reached and or the final discontinuation of the treatment
Temporary discontinuation of treatment with Saizen if > 1 week (number, duration, person responsible for the discontinuation, reason, dose upon resumption of treatment) and final discontinuation of treatment with Saizen (date and reason) | Inclusion visit to follow-up visits at 3, 6 and 12 month and annual until the adult height is reached and or the final discontinuation of the treatment
Biochemical and endocrinological parameters | Inclusion visit to follow-up visits at 3, 6 and 12 month and annual until the adult height is reached and or the final discontinuation of the treatment
  * Tolerance
  * Concomitant treatments

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Chatelain, MD, Professor, Study Chair — Service d'Endocrinologie Pédiatrique & Diabétologie Infantile, Hôpital Femme Mère Enfant, Lyon-Bron, France
Locations (40):
- France (40):
  - Merck Serono Investigational Site, Aix-en-Provence
  - Merck Serono Investigational Site, Annemasse
  - Merck Serono Investigational Site, Belfort
  - Merck Serono Investigational Site, Besançon
  - Merck Serono Investigational Site, Bordeaux
  - Merck Serono Investigational Site, Brest
  - Merck Serono Investigational Site, Caen
  - Merck Serono Investigational Site, Chambéry
  - Merck Serono Investigational Site, Clermont-Ferrand
  - Merck Serono Investigational Site, Dijon
  - Merck Serono Investigational Site, Fréjus
  - Merck Serono Investigational Site, Grenoble
  - Merck Serono Investigational Site, Hyères
  - Merck Serono Investigational Site, La Rochelle
  - Merck Serono Investigational Site, Laon
  - Merck Serono Investigational Site, Le Havre
  - Merck Serono Investigational Site, Le Mans
  - Merck Serono Investigational Site, Lille
  - Merck Serono Investigational Site, Limoges
  - Merck Serono Investigational Site, Lisieux
  - Merck Serono Investigational Site, Ludres
  - Merck Serono Investigational Site, Lyon-Bron
  - Merck Serono Investigational Site, Marseille
  - Merck Serono Investigational Site, Mâcon
  - Merck Serono Investigational Site, Montbéliard
  - Merck Serono Investigational Site, Montluçon
  - Merck Serono Investigational Site, Montpellier
  - Merck Serono Investigational Site, Nantes
  - Merck Serono Investigational Site, Nice
  - Merck Serono Investigational Site, Orléans
  - Merck Serono Investigational Site, Paris
  - Merck Serono Investigational Site, Pringy
  - Merck Serono Investigational Site, Puyricard
  - Merck Serono Investigational Site, Reims
  - Merck Serono Investigational Site, Saint-Priest-en-Jarez
  - Merck Serono Investigational Site, Strasbourg
  - Merck Serono Investigational Site, Toulon
  - Merck Serono Investigational Site, Toulouse
  - Merck Serono Investigational Site, Tours
  - Merck Serono Investigational Site, Vesoul